CLINICAL TRIAL: NCT01312649
Title: Feeling of Being in Control of One's Own Action: Which Mechanisms in Healthy Volunteers and in Mental Diseases
Brief Title: Feeling of Being in Control of One's Own Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 4880
Record Dates: First submitted 2011-03-01; First posted 2011-03-11 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Bipolar Disorders
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental): Healthy volunteers
  Interventions: Behavioral: Experimental psychology methods (computer tests)
- Arm 2 (Experimental): Schizophrenia with history of delusions of control
  Interventions: Behavioral: Experimental psychology methods (computer tests)
- Arm 3 (Experimental): Schizophrenia without history of delusions of control
  Interventions: Behavioral: Experimental psychology methods (computer tests)
- Arm 4 (Experimental): Bipolar disorders
  Interventions: Behavioral: Experimental psychology methods (computer tests)
- Arm 5 (Active Comparator): Matched healthy controls
  Interventions: Behavioral: Experimental psychology methods (computer tests)

INTERVENTIONS:
Behavioral: Experimental psychology methods (computer tests)

SUMMARY:
The investigators aim is to understand the cognitive mechanisms that contribute to the emergence of delusions of control (the belief that one's own actions or thoughts are controlled by an external force). These symptoms are mainly encountered in patients with schizophrenia, and the investigators will distinguish patients with schizophrenia with or without this symptom together with patients with bipolar disorder. Based on the investigators previous studies, this project will help to determine the role of two elementary mechanisms in the ability to feel in control of voluntary actions: (1) the processing of the sensory consequences of action, and (2) the ability to build mental representations for sequenced actions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia or bipolar disorders (criteria DSM IV) or healthy controls matched with patients on age, sex and education level
* 18-55 years old

Exclusion Criteria:

* Past history affecting CNS
* Invalidating sensory disorders
* Intake of psychotropic drugs, except for patients
* Intake of benzodiazepines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne GIERSCH, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Pôle de Psychiatrie - Hôpital civil, Strasbourg, France

REFERENCES:
- [Result] Turgeon M, Giersch A, Delevoye-Turrell Y, Wing AM. Impaired predictive timing with spared time interval production in individual with schizophrenia. Psychiatry Res. 2012 May 15;197(1-2):13-8. doi: 10.1016/j.psychres.2012.03.003. Epub 2012 Apr 11. PMID 22497958